CLINICAL TRIAL: NCT02055001
Title: Haemostasis Evaluation Related to Sexual Hormones: Gender Perspective
Brief Title: Sexual Hormones and Haemostasis: Observations for Women Health
Acronym: SHOW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Stefania Basili, Prof., University of Roma La Sapienza
Other Study IDs: SHOW
Record Dates: First submitted 2014-01-20; First posted 2014-02-04 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Gender; Sex
Keywords: gender medicine; platelet function; sex hormones; antiplatelet drugs; haemostasis
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum samples Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Atherothrombotic disorders account for 25% of all deaths among women and for substantial morbidity and resource use in health care. Nonetheless, gender-related differences in the epidemiology of cardiovascular disease (CVD) remain largely unexplained. Among mechanisms that could account for such differences, the biology of platelets, which exert a pivotal pathogenetic role in atherothrombosis, and of coagulation system are on investigation.

Thus, differences in platelet reactivity between women and men have been described using several methods and in response to varying stimuli. Indeed, sex steroid hormones could be involved in a different response of platelet to physiological response to agonists. The finding that estrogen receptors are expressed in platelets makes these cells an excellent model for studying the non-genomic effects of steroid hormones. Also coagulation cascade has been reported to be influenced by sexual endogenous as well as exogeneous hormones (i.e contraceptives) In particular, the impact of endogenous estrogens (menstrual cycle) on platelet activity and on response to antiplatelets drugs in fertile women has never been evaluated.

Accordingly, the goal of this proposal is to investigate relationship between platelet function (assessed by aggregometry tests and markers of platelet activation in vivo such as thromboxane production, CD40L and P- selectin levels) and sex hormones during physiological regular menstrual cycles (28-30 days) in healthy pre-menopausal women aged from 18 to 40 years. Moreover, in a subgroup of healthy women free from antiplatelet drugs, will be planned a proof of concept study to investigate if there will be variations, during a short term (1 month) low dose aspirin, in platelet reactivity according to the different phases of menstrual cycle in 10 healthy premenopausal women aged from 18 to 40 years. Moreover, it will be investigate effect of steroid hormonal pattern on residual platelet activity response on treatment

DETAILED DESCRIPTION:
Atherothrombotic disorders account for 25% of all deaths among women and for substantial morbidity and resource use in health care. Nonetheless, gender-related differences in the epidemiology of cardiovascular disease (CVD) remain largely unexplained. Thus, the application of sex-gender medicine is strongly recommended by WHO and other international organization. In fact, it is emerging that although men and women are subject to the same cardiovascular diseases (CVD), however, they have different risk factors, disease progression and response to drug treatment.

In the last decades emerging scientific knowledge about platelet role in the atherothrombotic diseases physiopathology provides clues and asks questions about the possibility that a different platelet function modulation could influence the women population cardiovascular disease clinical course, especially considering that, compared to men population, the women one recognizes a worst cardiovascular outcome.

It is widely acknowledged that platelet reactivity plays a pivotal role in thrombus formation and atherosclerosis. Differences in platelet reactivity between women and men have been described using several methods and in response to varying stimuli. In particular, platelets from women without vascular diseases are more reactive than those of men in response to standard concentrations of agonists such as adenosine diphosphate (ADP) and thrombin receptor agonist protein. Mechanisms that could account for such differences are on investigation. Indeed, sex steroid hormones could be involved as they exert multiple direct and indirect effects on cardiovascular physiology. The pleiotropic effects of estradiol-17 (E2) and estrogen receptors (ERs), a part of thei pivotal role in sexual development and reproduction,are a consequence of both the widespread expression of ER in many cell populations within the body as well as possibly reflecting the ancestral status of ER in the steroid receptor family.

Epidemiologic and experimental studies now support an atheroprotective effect of both endogenous and exogenous estrogens. The Women's Health Initiative study did not show a coronary protective effect of estrogen in postmenopausal women, but subsequent studies have shown that this was because of both inappropriate timing (ie, administering the hormone therapy too late) and the identity of the associated progestin.

Physiologic differences between men and women affect also drug activity, including pharmacokinetics and pharmacodynamics. Women are underrepresented in cardiovascular studies, even as their preponderance in the aging population steadily increases. A better understanding of the factors contributing to the observed sex-related differences in platelet biology is warranted. In particular concerns have been raised about the role of specific hormones in mediating platelet activation and function and the differential benefit of antiplatelet medications for women.

It has been reported that many of sex gender differences associated with CVD in women could depend by estrogen. The finding that estrogen receptors are expressed in platelets renders these cells an excellent model for studying the non-genomic effects of these hormones.

In conclusion, the impact of estrogens endogenous (menstrual cycle) and/or exogenous (oral contraceptives therapy) on platelet activity and response to antiplatelets drugs in women has not been extensively evaluated.

To fill this gap in evidence and to find a support to optimize cardiovascular therapy by gender-oriented approach, the investigators planned to study the effect of endogenous estrogens (menstrual cycle) on platelet function and on antiplatelet therapy response in pre-menopausal healthy women.

Phase 1 Evaluation of platelet function in different menstrual cycle phases. Phase 2: "Proof of concept study" A short treatment period with aspirin (100 mg daily) was also planned. Patients involved in the first phase study will be asked to participate in the interventional study. The investigators plan to enroll in the study 10 women and to follow them for 1 month.

Blood samples will be obtained at baselines and at four time points during treatment to verify the effect of aspirin on platelets' function related to menstrual cycle hormonal fluctuations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pre-menopausal women wiith regular menstrual cycle
* Age 18 - 40 years
* Written Informed Consent

Exclusion Criteria:

* History of recent (within the last 2 months) ingestion of anticoagulants, antifibrinolytics, non-steroidal antiinflammatory medications, combined oral contraceptives, and progestagens.
* Pregnancy
* Presence of kidney, liver, heart, endocrine diseases or infective diseases for at least 2 months prior to the study
* No history of gastrointestinal disease at risk of bleeding and/or previous gastrointestinal bleeding
* Use chronic pharmaceutical treatments

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 21 healthy women with 28-30 day regular menstrual cycle
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in platelet activation markers levels according to sex hormones levels at the beginnig, during and at the end of a physiological regular menstrual cycles (28-30 days) in healthy pre-menopausal women. | baseline (beginning of menstruation); day 5 ± 2; day 14 ± 2; day 21 of menstrual cycle, according to the hormonal fluctuations
  To investigate relationship between platelet function (assessed by aggregometry tests and markers of platelet activation in vivo such as thromboxane production, CD40L and P- selectin levels) and sex hormones during physiological regular menstrual cycles (28-30 days) in healthy pre-menopausal women aged from 18 to 40 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Basili, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome - Policlinico Umberto I Roma, Rome, I, Italy